CLINICAL TRIAL: NCT07086846
Title: Effect of Myofascial Release Versus Acupressure on Carpal Tunnel Syndrome in Postnatal Period
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Kamal Abd El-Aal Mansour, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/005373
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Myofascial Release Therapy; Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release technique (Experimental): The participants will receive myofascial release, for 15 minutes, three times per week for 6 weeks (total of 18 sessions), in addition to night splint and home advice.
  Interventions: Other: Night splint; Other: Myofascial release technique; Other: Home advice
- Acupressure (Experimental): The participants will receive acupressure on pericardium 6 acupoint (PC-6 point) for 3 minutes, three times per week for 6 weeks (total of 18 sessions), in addition to night splint and home advice.
  Interventions: Other: Night splint; Other: Acupressure; Other: Home advice

INTERVENTIONS:
Other: Night splint — All participants will be treated conservatively by wrist splint in a neutral position.
Other: Myofascial release technique — The participant will receive myofascial release using M2T blade. It will be applied on the carpal tunnel over and above the wrist creases on the ventral aspect of the forearm for 15 minutes, 3 sessions weekly for 6 weeks (total of 18 sessions).
  Arms: Myofascial release technique
Other: Acupressure — It will be applied on the pericardium 6 point (PC-6) for 3 minutes, three times per week for 6 weeks (total of 18 sessions).
  It is located on the palm side of the wrist a couple of inches toward the body in between the two tendons (palmaris longus & flexor carpi radialis) that run approximately down the center of the forearm.
  Arms: Acupressure
Other: Home advice — The participants will be asked to follow important advices like supporting the wrists during activity and ensuring proper posture, avoiding wrist flexion and extension, avoiding hard clutches, holding or carrying objects for a long time, catching with fingers, repetitive hand and wrist movement such as knitting or sewing, driving, activities and hobbies such as golf, tennis, table tennis.

SUMMARY:
This study will be conducted to compare the effect of myofascial release and acupressure on postnatal carpal tunnel syndrome.

DETAILED DESCRIPTION:
Various factors, such as an increase in body mass index (BMI), hormones (relaxin), fluid redistribution, and maternal age, are involved in the etiology of pregnancy related carpal tunnel syndrome (CTS). In terms of prognosis, although it has been reported that pregnancy related CTS generally regresses completely spontaneously or with conservative treatment methods after birth, residual symptoms and neurophysiological findings that require surgical decompression up to a year after birth have also been reported.

In clinical practice guidelines, conservative treatment is recommended for mild and moderate cases, while a surgical approach is recommended for patients with severe CTS . Some clinical conditions such as hormonal alteration and edema for menopause and pregnancy due to alteration of the fluid balance in the body.

Myofascial release is considered a safe, non-invasive, and simple method for decreasing pain intensity and numbness sensation severity and for improving hand function in pregnant women with CTS.

Acupressure is the supportive therapies based on Chinese medicine. Pressure is applied to the affected areas without the use of needles. PC7 or the Daling point is especially considered when managing CTS; it was found to cause an increase of endomorpin-1, beta-endorphin, serotonin, dopamine, and enkephalin levels in the brain tissues and plasma. Acupressure was found to be more effective compared to the placebo and splints re- garding the functional status and nerve conduction studies.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women with mild to moderate carpal tunnel syndrome (CTS).
* Their ages will range from 25 to 35 years old.
* Their body mass index (BMI) will range from 25 to 30 Kg/m2.
* The electrophysiological evidence of mild or moderate median nerve lesion at wrist (mild: sensory nerve conduction velocity slow on finger/wrist measurement, sensory nerve latency >3.5 ms, normal terminal motor latency; moderate: sensory potential preserved with motor slowing, distal motor latency to abductor pollicis brevis (APB) < 6.5 ms)
* Positive phalen's test.
* Positive tinel's test.
* Unilateral or bilateral carpal tunnel affection will be included.

Exclusion Criteria:

* History of brachial plexopathy or malignancy.
* Radial, ulnar neuropathy, proximal median neuropathy or polyneuropathy.
* Previous wrist surgery or steroid injection for CTS.
* History of trauma, fracture, deformity or inflammation in the wrist, such as rheumatoid arthritis.
* Coagulation abnormalities, pregnancy, fever and infections.
* Skin disease and skin cancer.
* Spots, birthmarks or tattoos over the work points.
* Pacemaker and implementable medical devices.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-07-27 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 6 weeks
  The visual analogue scale (VAS) will be used to assess pain intensity before and after intervention. The VAS is usually presented as a 10-cm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
Sensory conduction velocity | 6 weeks
  Electromyography device (Tru Trace EMG, 2ch Head box device, manufactured by deymed Diagnostic Pvt., Ltd., Czech Republ) will be used to assess sensory conduction velocity of median nerve before and after the treatment. A pair of ring electrodes will be placed on the index finger for recording, and the sensory nerve will be stimulated antidromically. The stimulating electrodes will be placed at the wrist proximal to carpal tunnel for the distal segment stimulation and at the elbow medial to biceps tendon for the proximal segment stimulation.
  Conduction velocity is the speed at which the electrical signal travels along the nerve. A reduced velocity can also indicate nerve damage. Its normal range is from 44-60 ms.
Sensory distal latency | 6 weeks
  Electromyography device (Tru Trace EMG, 2ch Head box device, manufactured by deymed Diagnostic Pvt., Ltd., Czech Republ) will be used to assess sensory distal latency of median nerve before and after the treatment. A pair of ring electrodes will be placed on the index finger for recording, and the sensory nerve will be stimulated antidromically. The stimulating electrodes will be placed at the wrist proximal to carpal tunnel for the distal segment stimulation and at the elbow medial to biceps tendon for the proximal segment stimulation. The distal motor latency is measured from the onset of the stimulating artifact to the onset of the compound muscle action potential. Its normal range is from 2.5-3.5 ms.
Median nerve amplitude | 6 weeks
  The amplitude of the median nerve (specifically, the sensory nerve action potential, or SNAP) will be measured by electromyography (Tru Trace EMG, 2ch Head box device, manufactured by deymed Diagnostic Pvt., Ltd., Czech Republ) during nerve conduction study before and after treatment. It is measured in microvolts (µV) and reflects the number of nerve fibers conducting the electrical signal. During a nerve conduction study, a small electrical stimulus is applied to the median nerve, and the resulting electrical activity is recorded. The amplitude is then measured as the height of the waveform generated by this activity. Its normal value should be at least 6 microvolt (6 µV).

SECONDARY OUTCOMES:
Assessment of severity of carpal tunnel syndrome symptoms | 6 weeks
  Boston Carpal Tunnel Questionnaire will be used before and after intervention. It comprises two scales, a symptom severity scale (SSS) and a functional status scale (FSS). The SSS evaluates symptoms with regard to severity, frequency, and time. The FSS indicates how the syndrome affects daily life. SSS involves 11 questions, addressing: pain intensity during day time and night time, time of pain during the day, numbness, weakness, tingling sensation at night, frequency of night tingling sensation, and skill. Each question offers 5 answers, from 0 points (no symptoms) to 4 points (most severe symptoms). Questions concerning FSS refer to daily activities that will be performed by most individuals and are commonly affected by CTS. The patients rate their ability to perform each activity on a scale that ranged from 1 point (no difficulty with the activity) to 5 points (cannot perform the activity at all).The overall score for the FSS is the mean of the ratings on the daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Botla, Professor, Study Director — Cairo University; Soheir El-kosery, Professor, Study Chair — Cairo University
Locations (1):
- Amr Kamal Abd El-Aal, Cairo, Egypt